CLINICAL TRIAL: NCT03687957
Title: Effect of rhIL-7-hyFc on Increasing Lymphocyte Counts in Patients With Newly Diagnosed Non-severe Lymphopenic Gliomas Following Radiation and Temozolomide
Brief Title: rhIL-7-hyFc on Increasing Lymphocyte Counts in Patients With Newly Diagnosed Non-severe Lymphopenic Gliomas Following Radiation and Temozolomide
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: NeoImmuneTech (Industry); The Foundation for Barnes-Jewish Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 201810185
Record Dates: First submitted 2018-09-25; First posted 2018-09-27 (Actual); Results first posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — efineptakin alfa; Temozolomide; Radiotherapy

STUDY DESIGN:
Intervention Model Description: -Phase I enrollment will be a sequential enrollment (patients will be stratified by concomitant use of steroids (yes/no). Phase II randomized portion will open with 2 arms being enrolled to in parallel. Phase II expansion cohort will not be randomized.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Phase II only: This study is triple-blinded (participant, physician, and study coordinator are all blinded; pharmacist and study statistician are not blinded)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (9):
- Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) (Experimental): * Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 7 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned
  * The phase I part will begin with an Accelerated Phase with 1 patient per cohort at the first 2 doses (60 mcg/kg and 120 mcg/kg) followed by a standard 3+3 design on the remaining 4 dose levels
  Interventions: Drug: rhIL-7-hyFc; Drug: Temozolomide; Radiation: Radiation therapy
- Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) (Experimental): * Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 7 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned
  * The phase I part will begin with an Accelerated Phase with 1 patient per cohort at the first 2 doses (60 mcg/kg and 120 mcg/kg) followed by a standard 3+3 design on the remaining 4 dose levels
  Interventions: Drug: rhIL-7-hyFc; Drug: Temozolomide; Radiation: Radiation therapy
- Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) (Experimental): * Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 7 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned
  * The phase I part will begin with an Accelerated Phase with 1 patient per cohort at the first 2 doses (60 mcg/kg and 120 mcg/kg) followed by a standard 3+3 design on the remaining 4 dose levels
  Interventions: Drug: rhIL-7-hyFc; Drug: Temozolomide; Radiation: Radiation therapy
- Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) (Experimental): * Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 7 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned
  * The phase I part will begin with an Accelerated Phase with 1 patient per cohort at the first 2 doses (60 mcg/kg and 120 mcg/kg) followed by a standard 3+3 design on the remaining 4 dose levels
  Interventions: Drug: rhIL-7-hyFc; Drug: Temozolomide; Radiation: Radiation therapy
- Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) (Experimental): * Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 7 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned
  * The phase I part will begin with an Accelerated Phase with 1 patient per cohort at the first 2 doses (60 mcg/kg and 120 mcg/kg) followed by a standard 3+3 design on the remaining 4 dose levels
  Interventions: Drug: rhIL-7-hyFc; Drug: Temozolomide; Radiation: Radiation therapy
- Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) (Experimental): * Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 7 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned
  * The phase I part will begin with an Accelerated Phase with 1 patient per cohort at the first 2 doses (60 mcg/kg and 120 mcg/kg) followed by a standard 3+3 design on the remaining 4 dose levels
  Interventions: Drug: rhIL-7-hyFc; Drug: Temozolomide; Radiation: Radiation therapy
- Randomized Phase II: Placebo (Experimental): -Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. Placebo will be given by intramuscular injection starting at the end of RT/TMZ (within 14 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of placebo injections are planned.
  Interventions: Drug: Placebo; Drug: Temozolomide; Radiation: Radiation therapy
- Randomized Phase II: rhIL-7-hyFc (Experimental): Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 14 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned.
  Interventions: Drug: rhIL-7-hyFc; Drug: Temozolomide; Radiation: Radiation therapy
- Phase II Expansion Arm: rhIL-7-hyFc (Experimental): Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 14 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned.
  Interventions: Drug: rhIL-7-hyFc; Drug: Temozolomide; Radiation: Radiation therapy

INTERVENTIONS:
Drug: rhIL-7-hyFc — -Given by intramuscular injection
  Arms: Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg); Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg); Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg); Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg); Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg); Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg); Phase II Expansion Arm: rhIL-7-hyFc; Randomized Phase II: rhIL-7-hyFc
Drug: Placebo — -Given by intramuscular injection
  Arms: Randomized Phase II: Placebo
Drug: Temozolomide — -Standard of care
  Other Names: TMZ
Radiation: Radiation therapy — -Standard of care
  Other Names: RT

SUMMARY:
The investigators have developed a phase I/II clinical trial to evaluate the effect of rhIL-7-hyFc on lymphocyte counts in patients with high grade glioma (HGG).

A phase I study will test whether rhIL-7-hyFc can be safely administered to patients with HGG. Six doses of rhIL-7-hyFc will be tested using a mix of Accelerated Phase and standard 3+3 dose-escalation design. The phase II portion to test effect of rhIL-7-hyFc on lymphocyte counts will use placebo-controlled randomization in HGG patients whose treatment include the standard radiation therapy (RT) and temozolomide (TMZ).

ELIGIBILITY:
Inclusion Criteria:

* World Health Organization (WHO) grade III, grade IV, and high risk grade II gliomas that require RT and TMZ treatment.
* Phase 2 Expansion Cohort ONLY: Must be IDH1 wildtype, as defined by negative immunohistochemistry using an R132H-specific antibody and MGMT promoter unmethylated glioblastoma multiforme (WHO grade IV).
* Post-operative treatment must have included radiation and TMZ. Prior Gliadel Wafers are allowed. Glucocorticoid therapy is allowed. Tumor treating fields (TTF) device is allowed.
* Adequate organ and marrow function defined as follows:

  * Absolute neutrophil count ≥ 1,000/mcL
  * Platelets ≥ 75,000/mcL
  * Hemoglobin ≥ 8 g/dL
  * Total bilirubin ≤ 3.0 x institutional upper limit of normal
  * AST (SGOT)/ALT (SGPT) ≤ 3.0 × institutional upper limit of normal
  * Absolute lymphocyte count (ALC) ≥ 600/mcL (required for phase I and randomized phase II only)
* Karnofsky Performance Status (KPS) ≥ 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Able to provide written informed consent (or consent from a legally authorized representative).
* Women of childbearing potential must have a negative serum pregnancy test prior to study entry (within 14 days). Patients must be willing to be on adequate contraception during treatment.

  * 18 years of age.

Exclusion Criteria:

* Receiving any other investigational agents which may affect patient's lymphocyte counts.
* Pregnant women are excluded from this study because rhIL-7-hyFc has not been evaluated regarding its potential for teratogenic or abortifacients effects. There is a potential risk for adverse events in nursing infants secondary to treatment of the mother with the study drug, breastfeeding should be discontinued if the mother is treated with rhIL-7-hyFc.
* Has an active viral infection requiring systemic treatment at screening.
* Has active autoimmune disease or syndrome (i.e. moderate or severe rheumatoid arthritis, moderate or severe psoriasis, multiple sclerosis, myasthenia gravis, Guillain Barre syndrome, systemic lupus erythematosis, scleroderma, ulcerative colitis, Crohn's disease, autoimmune hepatitis, Wegener's etc.,) that requires systemic treatment at the time of screening. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment. Subjects are permitted to enroll if they have vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger.
* Receipt of live attenuated vaccine within 30 days before the first dose of study treatment. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, chicken pox, yellow fever, rabies, Bacillus Calmette-Guérin (BCG), Zoster, and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g. FluMist) are live attenuated vaccines and are not allowed.
* Has clinically significant cardiac enzymes ([Tnl or TnT] or CK-MD)
* Patients with a clinically significant EKG on screening triggering a echocardiogram which is also clinically significant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2028-04-13 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Milan Chheda, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Campian JL, Ghosh S, Kapoor V, Yan R, Thotala S, Jash A, Hu T, Mahadevan A, Rifai K, Page L, Lee BH, Ferrando-Martinez S, Wolfarth AA, Yang SH, Hallahan D, Chheda MG, Thotala D. Long-Acting Recombinant Human Interleukin-7, NT-I7, Increases Cytotoxic CD8 T Cells and Enhances Survival in Mouse Glioma Models. Clin Cancer Res. 2022 Mar 15;28(6):1229-1239. doi: 10.1158/1078-0432.CCR-21-0947. PMID 35031547
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The Phase II Expansion Arm never opened to enrollment and no participants were enrolled in this portion of the trial.
Groups:
- Randomized Phase II: Not Randomized: Enrolled to Randomized Phase II trial portion but not randomized.
Period: Overall Study
Arm/Group | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) | Randomized Phase II: Placebo | Randomized Phase II: rhIL-7-hyFc | Randomized Phase II: Not Randomized | Phase II Expansion Arm: rhIL-7-hyFc
Started | 1 | 1 | 3 | 6 | 6 | 2 | 11 | 11 | 1 | 0
Completed | 1 | 0 | 2 | 0 | 2 | 0 | 4 | 5 | 0 | 0
Not Completed | 0 | 1 | 1 | 6 | 4 | 2 | 7 | 6 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 1 | 0
Not completed — Disease progression | 0 | 1 | 1 | 2 | 2 | 0 | 2 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0 | 0
Not completed — New malignancy | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 0
Not completed — Patient went on hospice | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) | Randomized Phase II: Placebo | Randomized Phase II: rhIL-7-hyFc | Randomized Phase II: Not Randomized | Total
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6 | 2 | 11 | 11 | 1 | 42
Age, Continuous [Median (Full Range); unit: years] | 57 [57 to 57] | 32 [32 to 32] | 46 [45 to 66] | 63 [24 to 67] | 57.5 [30 to 77] | 34 [30 to 38] | 58 [33 to 74] | 61 [44 to 74] | 42 [42 to 42] | 57.5 [24 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 3 | 1 | 5 | 4 | 1 | 15
  Male | 1 | 1 | 3 | 5 | 3 | 1 | 6 | 7 | 0 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 1 | 3 | 6 | 5 | 2 | 11 | 11 | 1 | 41
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  White | 1 | 1 | 3 | 6 | 6 | 2 | 10 | 9 | 1 | 39
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 3 | 6 | 6 | 2 | 11 | 11 | 1 | 42

OUTCOME MEASURES:

1. Primary Outcome: Phase I Only: Safety and Tolerability of rhIL-7-hyFc as Measured by the Maximum Tolerated Dose (MTD) of rhIL-7-hyFc
Description: -The maximum tolerated dose (MTD) is defined as the dose level immediately below the non-tolerated dose. A total of at least 6 patients must be treated at a dose level for it to be considered the MTD.
Time Frame: Within 30 days of treatment start
Population: All Phase I participants are evaluable for this outcome measure.
Measure: Number; unit: mcg/kg
Groups:
- Phase I: rhIL-7-hyFc All Dose Levels: * Per standard treatment, patients will receive concurrent RT/TMZ followed by adjuvant TMZ on Days 1-5 of a 28-day cycle for a total of 6 cycles. rhIL-7hyFc will be given by intramuscular injection starting at the end of RT/TMZ (within 7 days after last day of RT/TMZ). The 2nd injection will be administered 3-5 days after the last dose of cycle 3 TMZ treatment (~week 13). The 3rd injection will be given 3-5 days after the last dose of cycle 6 TMZ treatment (~week 25). Note the 2nd and 3rd injections should be administered once between Day 3 through 5 following the last dose of TMZ to achieve the strongest response. The 4th injection (last injection in the study) will be given after completion of monthly TMZ (~Week 37). A total of 4 doses of rhIL-7-hyFc injections are planned
  * The phase I part will begin with an Accelerated Phase with 1 patient per cohort at the first 2 doses (60 mcg/kg and 120 mcg/kg) followed by a standard 3+3 design on the remaining 4 dose levels
Arm/Group | Phase I: rhIL-7-hyFc All Dose Levels
Number analyzed (Participants) | 19
mcg/kg | 720

2. Primary Outcome: Phase I: Safety and Tolerability of rhIL-7-hyFc as Measured by Number of Participants With Dose-limiting Toxicities (DLTs)
Description: -DLTs are defined in the protocol.
Time Frame: Within 30 days of treatment start
Population: This outcome measure is for Phase I participants only.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) | Randomized Phase II: Placebo | Randomized Phase II: rhIL-7-hyFc | Randomized Phase II: Not Randomized
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6 | 2 | 0 | 0 | 0
Participants | 0 | 0 | 0 | 0 | 0 | 2 |  |  |

3. Primary Outcome: Randomized Phase II: Percent Change in Absolute Lymphocyte Count (ALC)
Description: Absolute lymphocyte count (ALC) is a laboratory test that measures the exact number of lymphocytes in a microliter (µL) of blood. Lymphocytes are a type of white blood cell that play a crucial role in the immune system.
Time Frame: Baseline to Prior to adjuvant TMZ (approximately week 4)
Population: Only participants in the Randomized Phase II Placebo and Randomized Phase II rhIL-7-hyFc are evaluable for this outcome measure.
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) | Randomized Phase II: Placebo | Randomized Phase II: rhIL-7-hyFc | Randomized Phase II: Not Randomized
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 11 | 0
percent change |  |  |  |  |  |  | 16.66667 (28.36597) | 147.8261 (285.9597) |

4. Primary Outcome: Phase II Expansion Arm: Progression-free Survival (PFS)
Description: -Defined from date of surgery to date of progression or death due to disease or date of last clinical follow up.
Time Frame: Through completion of follow-up (estimated to be 5 years and 6 months)
Population: The Phase II Expansion Arm of the trial never opened to enrollment and no participants were enrolled.
Arm/Group | Phase II Expansion Arm: rhIL-7-hyFc
Number analyzed (Participants) | 0

5. Secondary Outcome: Phase I and Randomized Phase II: Immunogenicity as Measured by Anti-drug Antibodies (ADAs)
Description: * The formation of anti-drug antibodies (ADA) to rhIL-7-hyFc will be evaluated: BioAgilytix will perform both Elisa Binding (non-neutralizing) and neutralizing antibody assays according to their Standard Operating Procedure. The data will be presented if anti-drug antibodies are detected or not detected in the samples.
  * Week 1 will be prior to injection of 1st dose of rhIL-7-hyFc, week 13 will be prior to the 2nd dose of rhIL-7-hyFc, and week 45 will be 8 weeks after the last dose of rhIL-7-hyFc.
Time Frame: Week 1, Week 13, Week 25, and Week 45
Population: Samples were not collected at all time points if a participant was removed from treatment or removed from the study prior to that timepoint. Week 25 was removed with amendment #4 and only one participant had a sample collected at this time point.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) | Randomized Phase II: Placebo | Randomized Phase II: rhIL-7-hyFc | Randomized Phase II: Not Randomized
Number analyzed (Participants) | 1 | 1 | 3 | 6 | 6 | 2 | 11 | 11 | 0
Participants
  Week 1: Detected | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 |
  Week 1: Not Detected | 1 | 1 | 3 | 6 | 5 | 2 | 9 | 10 |
  Week 13: number analyzed (Participants) | 1 | 1 | 3 | 2 | 5 | 0 | 7 | 7 | 0
  Week 13: Detected | 1 | 1 | 2 | 2 | 5 | 0 | 1 | 7 |
  Week 13: Not Detected | 0 | 0 | 1 | 0 | 0 | 0 | 6 | 0 |
  Week 25: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Week 25: Detected | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Week 25: Not Detected | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |
  Week 45: number analyzed (Participants) | 1 | 0 | 2 | 0 | 1 | 0 | 4 | 5 | 0
  Week 45: Detected | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 5 |
  Week 45: Not Detected | 0 | 0 | 2 | 0 | 0 | 0 | 4 | 0 |

6. Secondary Outcome: Phase I: Percent Change in Absolute Lymphocyte Count (ALC)
Description: as for outcome 3
Time Frame: Baseline to Prior to adjuvant TMZ (approximately week 4)
Population: Only Phase I participants are evaluable for this outcome measure.
Measure: Median (Standard Deviation); unit: percent change
Arm/Group | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) | Randomized Phase II: Placebo | Randomized Phase II: rhIL-7-hyFc | Randomized Phase II: Not Randomized
Number analyzed (Participants) | 1 | 1 | 3 | 3 | 6 | 2 | 0 | 0 | 0
percent change | 37.5 (NA) — SD was not able to be calculated because data is for 1 participant | -22.222 (NA) — SD was not able to be calculated because data is for 1 participant | 25 (161.231) | 129.545 (81.696) | 52.083 (87.525) | -5.639 (88.787) |  |  |

ADVERSE EVENTS:
Time Frame: - Serious adverse events and adverse events were collected from start of treatment through 30 days after end of treatment (median length of follow-up 215 days, full length 28-493 days). - All cause mortality is collected from enrollment date until 5 years following end of study treatment (median length of follow-up 561.5 days, full length 1-2271 days). 5 participants are still in follow-up for all-cause mortality.
Arm/Group | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) | Randomized Phase II: Placebo | Randomized Phase II: rhIL-7-hyFc | Randomized Phase II: Not Randomized
All-Cause Mortality (participants affected / at risk) | 1/1 | 1/1 | 1/3 | 5/6 | 5/6 | 2/2 | 9/11 | 10/11 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 0/3 | 2/6 | 4/6 | 1/2 | 3/11 | 4/11 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 3/3 | 5/6 | 6/6 | 2/2 | 9/11 | 11/11 | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) (N=1) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) (N=1) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) (N=3) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) (N=6) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) (N=6) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) (N=2) | Randomized Phase II: Placebo (N=11) | Randomized Phase II: rhIL-7-hyFc (N=11) | Randomized Phase II: Not Randomized (N=1)
Heart failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Fever (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA
Suspected neoplasm progression (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA
COVID-19 infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Car accident injuries (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Muscle weakness right-sided (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Seizure (Nervous system disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | NA
Stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I: rhIL-7-hyFc Dose Level 1 (60 mcg/kg) (N=1) | Phase I: rhIL-7-hyFc Dose Level 2 (120 mcg/kg) (N=1) | Phase I: rhIL-7-hyFc Dose Level 3 (240 mcg/kg) (N=3) | Phase I: rhIL-7-hyFc Dose Level 4 (540 mcg/kg) (N=6) | Phase I: rhIL-7-hyFc Dose Level 5 (720 mcg/kg) (N=6) | Phase I: rhIL-7-hyFc Dose Level 6 (960 mcg/kg) (N=2) | Randomized Phase II: Placebo (N=11) | Randomized Phase II: rhIL-7-hyFc (N=11) | Randomized Phase II: Not Randomized (N=1)
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | NA
Hearing impaired (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 2 | NA
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | NA
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA
Chills (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | NA
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA
Fatigue (General disorders) | 1 | 0 | 0 | 1 | 1 | 0 | 3 | 2 | NA
Fever (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | NA
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 3 | NA
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Sinus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Tooth infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | NA
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | NA
CD4 lymphocytes decreased (Investigations) | 1 | 0 | 3 | 2 | 1 | 0 | 0 | 0 | NA
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1 | NA
White blood cell decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | NA
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | NA
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | NA
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 2 | NA
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | NA
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | NA
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | NA
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | NA
Tremors (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Renal calculi (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | NA
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | NA
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | NA
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | NA
Skin atrophy (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | NA
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | NA
Biopsy and Interstitial Laser Thermal Therapy (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | NA
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1 | 3 | 0 | 3 | 0 | NA
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | NA
Pain - starts in right foot and migrates to head (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Pain - right side (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | NA
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Muscle weakness - right-sided (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Seizure (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Altered mental status (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | NA

LIMITATIONS AND CAVEATS:
After completion of enrollment to the Phase I and Phase II Randomized portions of the trial, funding was depleted. Despite numerous attempts to gain new funding, the Phase II Expansion portion of the trial was never opened to enrollment. The results are late due to this reason.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/57/NCT03687957/Prot_SAP_000.pdf